CLINICAL TRIAL: NCT01190410
Title: An Open-label, Multicenter Study to Assess the Safety of Certolizumab Pegol in Children and Adolescents With Active Crohn's Disease Who Completed C87035 (NCT00899678) or Who Were Terminated From C87035
Brief Title: Extension Study to Assess Long Term Safety in Children and Adolescents With Crohn's Disease Receiving Certolizumab Pegol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR0012
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Crohn's Disease
Keywords: Certolizumab Pegol; Cimzia®; Crohn's Disease; Children and Adolescents with Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Certolizumab pegol: high-dose group (Experimental): 400 mg administered subcutaneously every 4 weeks for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  Interventions: Drug: certolizumab pegol
- Certolizumab pegol: low-dose group (weight adjusted) (Experimental): 200 mg administered subcutaneously every 4 weeks for subjects ≥ 40 kg or 100 mg for subjects 20 to < 40 kg
  Interventions: Drug: certolizumab pegol

INTERVENTIONS:
Drug: certolizumab pegol — 400 mg administered subcutaneously every 4 weeks for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg
  Other Names: Cimzia®; Crohn's Disease
  Arms: Certolizumab pegol: high-dose group
Drug: certolizumab pegol — 200 mg administered subcutaneously every 4 weeks for subjects ≥ 40 kg or 100 mg for subjects 20 to < 40 kg
  Other Names: Cimzia®; Crohn's Disease
  Arms: Certolizumab pegol: low-dose group (weight adjusted)

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of certolizumab pegol (CZP) treatment in children and adolescents with moderately to severely active Crohn's disease. Secondarily, to assess the long-term efficacy, pharmacokinetics (PK), and immunogenicity of CZP treatment in children and adolescents with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject who completed the C87035 study (NCT00899678) through Week 62 or assessments when their participation in C87035 was terminated when the study was stopped by UBC
* Subject completed all assessments required for Week 62/Visit 23 at the time of termination
* Subjects maintain stable regimen of concomitant medications for Crohn's Disease (CD) throughout study

Exclusion Criteria:

* Subject who did not complete the C87035 study (Week 62 Visit), was terminated or did not complete all of the Week 62 assessments when their participation from C87035 was terminated when the study was stopped by UCB but did not complete all assessments required for Week 62/Visit 23 at the time of termination

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877-822-9493 UCB
Locations (10):
- United States (7):
  - 114, Orange, California
  - 111, Aurora, Colorado
  - 103, Atlanta, Georgia
  - 116, Atlanta, Georgia
  - 112, Shreveport, Louisiana
  - 104, Baltimore, Maryland
  - 126, Morristown, New Jersey
- 301, Parkville, Victoria, Australia
- Canada (2):
  - 203, Edmonton, Alberta
  - 204, Hamilton, Ontario

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in August 2010 and concluded in November 2017.
Pre-assignment Details: The study included an Open Label treatment period, having 16 subjects enrolled in the Safety Set (SS) shown in the Participant Flow.
Groups:
- Certolizumab Pegol: Low-dose Group (Weight Adjusted): 200 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 100 mg for subjects 20 to < 40 kg. Part of the Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
- Certolizumab Pegol: High-dose Group (Weight Adjusted): 400 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 200 mg for subjects 20 to < 40 kg. Part of the Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
Period: Overall Study
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) | Certolizumab Pegol: High-dose Group (Weight Adjusted)
Started (16) | 4 | 12
Re-Induction | 0 | 2
Completed (6) | 3 | 3
Not Completed | 1 | 9
Not completed — Adverse Event | 0 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Administrative decision | 1 | 0
Not completed — PI discretion | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which included all subjects enrolled in the study.
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) | Certolizumab Pegol: High-dose Group (Weight Adjusted) | Total Title
Number analyzed (Participants) | 4 | 12 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 11 | 15
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.4) | 13.9 (2.9) | 13.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 3 | 3
  White | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least One Treatment-Emergent Adverse Event (TEAE) During Study Treatment (up to 303 Weeks)
Description: Treatment-Emergent Adverse Events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.
Time Frame: During study treatment (up to 303 weeks)
Population: The Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS): 200 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 100 mg for subjects 20 to < 40 kg. Part of the Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
- Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS): 400 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 200 mg for subjects 20 to < 40 kg. Part of the Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
- Certolizumab Pegol: Re-Induction Group - (SS): If a subject had not been previously reinduced in C87035, the subject is eligible for 1 reinduction due to loss of response in CR0012. Reinduction Week 0 (first reinduction dose) is followed by Reinduction Week 2 (second dose, 2 weeks after first dose), and Reinduction Week 4 (third dose, 2 weeks after second dose). The reinduction dose was adjusted to the subject's weight: 400 mg for subjects ≥ 40 kg or 200 mg for subjects 20 to < 40 kg subcutaneously Q2W for a total of 3 doses. After reinduction was complete participants continued dosing with CZP administered subcutaneously Q4W as 400 mg for subjects ≥ 40 kg or 200mg for subjects 20 to < 40 kg, regardless of the subject's previous randomized dose group). Part of the Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: Re-Induction Group - (SS)
Number analyzed (Participants) | 4 | 10 | 2
Participants
  Subjects | 2 | 6 | 2

2. Secondary Outcome: Number of Subjects Discontinuing Treatment Due to a Treatment-Emergent Adverse Event (TEAE)
Description: as for outcome 1
Time Frame: During study treatment (up to 303 weeks)
Population: The Safety Set (SS) included all subjects enrolled, who received at least 1 injection of study treatment in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: Re-Induction Group - (SS)
Number analyzed (Participants) | 4 | 10 | 2
Participants | 0 | 2 | 0

3. Secondary Outcome: Number of Subjects Who Develop Anti-nuclear Antibodies During the Study
Description: Anti-nuclear antibodies (ANA) are autoantibodies. ANA titers will be determined every 12 weeks starting at Week 14, and at the Completion/Early Termination and Safety Follow-Up (SFU) Visits.
Time Frame: At the time of completion or termination visit (up to 298 weeks)
Population: The Intention-to-Treat (ITT) Population included all subjects irrespective of any protocol deviations who received at least 1 injection of the study treatment and who had at least 1 efficacy measurement after the first injection of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (ITT): 200 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 100 mg for subjects 20 to < 40 kg. Part of the Intention-to-Treat (ITT) Population included all subjects irrespective of any protocol deviations who received at least 1 injection of the study treatment and who had at least 1 efficacy measurement after the first injection of this study.
- Certolizumab Pegol: High-dose Group (Weight Adjusted) - (ITT): 400 mg administered subcutaneously every 4 weeks for subjects >= 40 kg or 200 mg for subjects 20 to < 40 kg. Part of the Intention-to-Treat (ITT) Population included all subjects irrespective of any protocol deviations who received at least 1 injection of the study treatment and who had at least 1 efficacy measurement after the first injection of this study.
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (ITT) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (ITT)
Number analyzed (Participants) | 3 | 10
Participants | 0 | 3

4. Secondary Outcome: Number of Subjects Who Develop Double-stranded Deoxyribonucleic Acid (dsDNA) Antibodies During the Study
Description: Anti-dsDNA are autoantibodies. Anti-dsDNA titers will be determined every 12 weeks starting at Week 14, and at the Completion/Early Termination and Safety Follow-Up (SFU) Visits.
Time Frame: At the time of completion or termination visit (up to 298 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (ITT) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (ITT)
Number analyzed (Participants) | 3 | 10
Participants
  Subjects | 0 | 0

5. Secondary Outcome: Percentage of Subjects in Clinical Remission
Description: Percentage of subjects in clinical remission (clinical remission is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10)
Time Frame: At the time of completion or termination visit (up to 298 weeks)
Population: The Intention-to-Treat (ITT) Population included all subjects irrespective of any protocol deviations who received at least 1 injection of study treatment in this study and who had at least 1 efficacy measurement after the first injection of this study.
Measure: Number; unit: Percentage of particpiants
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (ITT) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (ITT)
Number analyzed (Participants) | 3 | 9
Percentage of particpiants | 100 | 44.4

ADVERSE EVENTS:
Time Frame: During study treatment (up to 303 weeks)
Arm/Group | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS) | Certolizumab Pegol: Re-Induction Group - (SS)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/10 | 1/2
Other Adverse Events (participants affected / at risk) | 2/4 | 5/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS) (N=4) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS) (N=10) | Certolizumab Pegol: Re-Induction Group - (SS) (N=2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol: Low-dose Group (Weight Adjusted) - (SS) (N=4) | Certolizumab Pegol: High-dose Group (Weight Adjusted) - (SS) (N=10) | Certolizumab Pegol: Re-Induction Group - (SS) (N=2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ultrasound abdomen (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (6) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2012-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT01190410/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT01190410/SAP_001.pdf